CLINICAL TRIAL: NCT02773043
Title: Evaluation of Myocardial Perfusion Reserve
Acronym: EVARESERVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC14.214
Record Dates: First submitted 2016-04-25; First posted 2016-05-16 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- non invasive imaging technique (Other)
  Interventions: Device: CZT SPECT camera

INTERVENTIONS:
Device: CZT SPECT camera

SUMMARY:
The proposed study is to validate a non-invasive imaging technique to evaluate the myocardial perfusion reserve in comparison with a validated invasive technique, the measure of coronary flow reserve (CRF) with thermodilution.

DETAILED DESCRIPTION:
Coronary artery disease is a public health problem. The measurement of myocardial perfusion reserve is a prognostic factor supplemental.

Its measure should influence the treatment and the follow up of the patients. The measurement of CRF by by one pressure-temperature sensor-tipped guide wire is a validated technique to evaluate the myocardial perfusion reserve but it is an invasive technique.

In this study, the investigators will compare this method with a non-invasive method: completely automated analysis and quantification of myocardial blood flow from DICOM files corresponding to stress and rest images was developed with a new camera CZT SPECT.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial scintigraphy with pharmacologic stress and abnormal results
* Coronarography indicated
* Informed consent

Exclusion Criteria:

* Pregnant woman
* Patient with terminal illness
* Terminal renal failure
* Allergy to iodine
* Informed consent impossible
* Patient under legal protection
* History of coronary artery bypass surgery
* Contraindications for adenosine: asthmatic patients, second or third-degree AV block without pacemaker or sick sinus syndrome. Systolic blood pressure less than 90 mmHg. Recent use of dipyramidole or dipyramidole-containing medications. Methyl xanthenes such as aminophylline caffeine or theobromine block the effect of adenosine and should be held for at least 12 hours prior to the test. Known hypersensitivity to adenosine. Unstable acute myocardial infarction or acute coronary syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Correlation between the measure of the coronary flow reserve with an invasive reference method (thermodilution) and a new non-invasive method in scintigraphy to measure the myocardial perfusion reserve | an average of 1 year
  Coronary flow reserve by thermodilution is the ratio between mean transit time of a room temperature 3-ml bolus of saline during rest and maximal hyperemia.
  Coronary flow reserve by CZT camera is given by ratio between Mycoardial perfusion during rest and maximal hyperemia. Myocardial perfusion is given by new software.

SECONDARY OUTCOMES:
Evaluation of the myocardial perfusion reserve measuring the CRF by thermodilution. | an average of 1 year
  Coronary flow reserve by thermodilution is the ratio between mean transit time of a room temperature 3-ml bolus of saline during rest and maximal hyperemia.
Evaluation of the myocardial perfusion reserve in scintigraphy by the same operator over different time scales and by two different operators. | an average of 1 year
  Coronary flow reserve by CZT camera is given by ratio between Mycoardial perfusion during rest and maximal hyperemia. Myocardial perfusion is given by new software.
Study the correlations between the level of soluble VE-cadherin (sVE) and the other indicators of coronary endothelial involvement (CRF and RMP). | Day of coronarography
  Blood test for soluble VE-cadherin (sVE), CRF, RMP

CONTACTS AND LOCATIONS:
Overall Officials: Gilles BARONE-ROCHETTE, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU Michallon, La Tronche, France

REFERENCES:
- [Result] Djaileb L, De Leiris N, Canu M, Sy OP, Seiller A, Leenhardt J, Charlon C, Faure M, Caillard J, Broisat A, Borel AL, Lablanche S, Betry C, Ghezzi C, Vanzetto G, Fagret D, Riou LM, Barone-Rochette G. Regional CZT myocardial perfusion reserve for the detection of territories with simultaneously impaired CFR and IMR in patients without obstructive coronary artery disease: a pilot study. J Nucl Cardiol. 2023 Aug;30(4):1656-1667. doi: 10.1007/s12350-023-03206-6. Epub 2023 Feb 22. PMID 36813934